CLINICAL TRIAL: NCT00621660
Title: Acupuncture Compared To Sham With a Placebo-Needle in Radiotherapy-Induced Nausea - a Randomised Controlled Study
Brief Title: Acupuncture Versus Sham for Radiotherapy-Induced Emesis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Linkoeping (Other)
Collaborators: Swedish Cancer Society (Other); Ostergotland County Council, Sweden (Other); Vardalinstitutet The Swedish Institute for Health Sciences (Other); Cancer & Traffic Injury Fund (Unknown)
Responsible Party: Senior Lecturer Sussanne Börjeson, Linkoeping University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 4960-B04-01XAC; 02-420; M167-04
Record Dates: First submitted 2008-02-11; First posted 2008-02-22 (Estimated); Last update posted 2008-02-22 (Estimated); Status verified 2007-11

CONDITIONS: Nausea; Vomiting
Keywords: Acupuncture therapy; Cancer; Emesis; Expectations; Placebo
MeSH Terms: conditions — Nausea; Vomiting; Neoplasms | interventions — Acupuncture Therapy; salicylhydroxamic acid

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Acupuncture (Experimental)
  Interventions: Procedure: Acupuncture
- Sham (Placebo Comparator)
  Interventions: Procedure: Sham

INTERVENTIONS:
Procedure: Acupuncture — Acupuncture was administered bilaterally to the standard antiemetic point2-4 pericardium six (PC6) located between the tendons of palmaris longus and flexor carpii radialis at two body-inches proximal of the wrist crease. Sharp needles, diameter 0.25 x length 40 millimetres, were inserted into a depth of a half body-inch. One body-inch (or a "cun" in traditional Chinese medicine context) is equivalent to the greatest width of the individual patients´ thumb at the distal phalanx, approximately one and a half centimetres or one American thumb. The needles were manipulated three times (at the start, middle and end of the treatment session) by twirling, thrusting and lifting until deqi occurred.
  Other Names: Invasive acupuncture
  Arms: Acupuncture
Procedure: Sham — Sham acupuncture was administered bilaterally to a non-acupuncture point two body-inches proximal of PC6 with the telescopic Park sham device16, 0.30 x 40 millimetres (fully extended length). That needle looks identical with a real needle but is blunted and glides upwards into its handle instead of penetrating, which gives an illusion of penetration. The marking tubes hold the needles in place. The therapist gave an illusion of manipulation by turning the needle three times, each time for a couple of seconds until the needle touched the skin, but no deqi occurred. Except when placing and manipulating the sham needle, it was not pressed against the skin at all.
  Other Names: Sham acupuncture; Placebo acupuncture
  Arms: Sham

SUMMARY:
The aim of this study is to evaluate if acupuncture prevents or reduces nausea or vomiting during radiotherapy

DETAILED DESCRIPTION:
Treatment with acupuncture is, despite sometimes unclear evidence, increasing in cancer care. Acupuncture is used for indications such as pain and nausea, but for radiotherapy (RT) induced nausea it is still an unexplored treatment. For evaluation of the method, the use of sham acupuncture as a control treatment provides a tool resembling placebo for drugs. The aim of the studt is therefore to investigate whether acupuncture reduces nausea caused by radiotherapy in a patient group with a >50% risk of experiencing the symptoms (abdominal or pelvic region). Patients are randomised to invasive acupuncture (IA) or placebo acupuncture (PA) 30 min, 2-3 times/week during the whole RT period. IA is administered bilaterally to the point PC6 using an invasive needle and PA with a needle, which looks identical but is not pointed and is not fixed in its handle. When this comes into contact with the surface of the skin and gives a feeling of penetration it glides upwards in its handle and is therefore shortened, which gives an illusion that the needle has entered the tissue. Nausea and vomiting is documented in diaries and questionnaires under the entire treatment period as well as two and four weeks after radiotherapy.

ELIGIBILITY:
Inclusion Criteria:

* patients of at least 18 years of age
* with gynaecologic-, anal-, rectal-, colon-, ventricle-, pancreatic- or testicular tumours
* willing to give their informed consent
* able to take part in the entire treatment and data collection procedure
* had planned radiation over an abdominal and/or pelvic field (with or without concomitant chemotherapy) with the volume of at least 800 cm3 and a dose of at least 25 Gy.

Exclusion Criteria:

* use of antiemetic treatment or persistent nausea within 24 hours prior to the start of radiotherapy
* ever received acupuncture against nausea, or during the last year received acupuncture for any indication.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 237 (Actual)
Dates: Start 2004-01; Primary Completion 2007-03 (Actual); Study Completion 2007-03 (Actual)

PRIMARY OUTCOMES:
Number of patients with at least one episode of nausea during the whole radiotherapy treatment period | The radiotherapy treatment period (md 5 weeks)

SECONDARY OUTCOMES:
Secondary outcome measures are the summed number of days with nausea, intensity of nausea, number of patients and summed number of days with vomiting, belief in the antiemetic effects and interest in receiving needling in the future | From acupunture start until 4 weeks after treatment stopped

CONTACTS AND LOCATIONS:
Overall Officials: Sussanne Börjeson, PhD, Principal Investigator — Linkoeping University
Locations (1):
- Sussanne Börjeson, Linköping, Sweden

REFERENCES:
- [Derived] Efverman A, Kristofferzon ML. A Basis for Strengthening Coping Strategies and Treatment Expectations in Patients Undergoing Emetogenic Pelvic-Abdominal Radiotherapy: A Longitudinal Study. Integr Cancer Ther. 2024 Jan-Dec;23:15347354241281329. doi: 10.1177/15347354241281329. PMID 39300870
- [Derived] Blom K, Efverman A. Sleep During Pelvic-Abdominal Radiotherapy for Cancer: A Longitudinal Study With Special Attention to Sleep in Relation to Nausea and Quality of Life. Cancer Nurs. 2021 Jul-Aug 01;44(4):333-344. doi: 10.1097/NCC.0000000000000826. PMID 32371667
- [Derived] Enblom A, Lekander M, Hammar M, Johnsson A, Onelov E, Ingvar M, Steineck G, Borjeson S. Getting the grip on nonspecific treatment effects: emesis in patients randomized to acupuncture or sham compared to patients receiving standard care. PLoS One. 2011 Mar 23;6(3):e14766. doi: 10.1371/journal.pone.0014766. PMID 21448267